CLINICAL TRIAL: NCT06944314
Title: Physicians' Perception About Patient Pain in Flexible Cystoscopy With Local Anesthesia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Associate Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MAR.UAD.0021
Record Dates: First submitted 2025-03-08; First posted 2025-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cystoscopic Surgical Procedures; Pain
Keywords: Pain; Anxiety; bladder cancer; Hematuria
MeSH Terms: conditions — Pain; Anxiety Disorders; Urinary Bladder Neoplasms; Hematuria | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The people who randomize the patient, prepare the patient for cystoscopy, perform the cystoscopy and evaluate the results are different and will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Assistant Urology Doctor (2 years) (Experimental): Intervention: Diagnostic Flexible Cystoscopy Other Names: Flexible Cystoscopy, Cystoscopy Arm Description: The procedure will be performed by an Assistant Urology Doctor with 2 years of experience. The goal is to evaluate the patient's pain perception during diagnostic flexible cystoscopy.
  Interventions: Procedure: Diagnostic procedures; Procedure: Flexible Cystoscopy
- Assistant Urology Doctor (4 years) (Experimental): Intervention: Diagnostic Flexible Cystoscopy Other Names: Flexible Cystoscopy, Cystoscopy Arm Description: The procedure will be performed by an Assistant Urology Doctor with 4 years of experience. The goal is to evaluate the patient's pain perception during diagnostic flexible cystoscopy.
  Interventions: Procedure: Diagnostic procedures; Procedure: Flexible Cystoscopy
- Specialist Urology Physician (<5 years experience) (Experimental): Experimental: Specialist Urology Physician (<5 years experience) Intervention: Diagnostic Flexible Cystoscopy Other Names: Flexible Cystoscopy, Cystoscopy Arm Description: The procedure will be performed by a Specialist Urology Physician with less than 5 years of experience. The goal is to evaluate the patient's pain perception during diagnostic flexible cystoscopy.
  Interventions: Procedure: Diagnostic procedures; Procedure: Flexible Cystoscopy
- Specialist Urology Physician (>5 years experience) (Experimental): Experimental: Specialist Urology Physician (>5 years experience) Intervention: Diagnostic Flexible Cystoscopy Other Names: Flexible Cystoscopy, Cystoscopy Arm Description: The procedure will be performed by a Specialist Urology Physician with more than 5 years of experience. The goal is to evaluate the patient's pain perception during diagnostic flexible cystoscopy.
  Interventions: Procedure: Diagnostic procedures; Procedure: Flexible Cystoscopy

INTERVENTIONS:
Procedure: Diagnostic procedures — Diagnostic Flexible Cystoscopy
  Other Names: Flexible Cystoscopy
Procedure: Flexible Cystoscopy — Diagnostic Flexible Cystoscopy
  Other Names: Cystoscopy

SUMMARY:
Cystoscopy with local anesthesia is commonly performed for the follow-up of bladder cancer, evaluation of hematuria, assessment of urethral strictures, and examination of the lower urinary tract. While some patients tolerate the procedure comfortably, others may exhibit heightened sensitivity and difficulty tolerating it. In certain cases, even when the procedure is completed, the level of pain experienced and the resistance demonstrated by the patient may render cystoscopy a challenging experience for both the patient and the physician. The physician's perception of the patient's pain may differ from the pain reported by the patient. Currently, there is no available data in the literature regarding the relationship between pre-procedural anxiety and depression levels and the pain experienced during cystoscopy, nor regarding the physician's perception of that pain. The primary objective of the study is to compare the patient-reported pain score with the physician's perception of the pain experienced by the patient. A secondary objective is to evaluate the pre-procedure anxiety and depression scores, along with intra-procedural pain scores, in patients undergoing flexible cystoscopy under local anesthesia.

DETAILED DESCRIPTION:
Cystoscopy is one of the most frequently performed procedures in the field of urology. Its widespread application, the impracticality of administering general anesthesia to all patients, and advancements in medical technology have led to the development of devices that enable cystoscopy to be performed with local or intraurethral anesthesia. As a result, cystoscopy under local anesthesia is commonly utilized for the follow-up of bladder cancer, evaluation of hematuria, assessment of urethral strictures, and examination of the lower urinary tract. Both rigid and flexible cystoscopes can be used for this purpose, with flexible instruments generally offering greater comfort for procedures involving local anesthesia.

In patients undergoing cystoscopy with local anesthesia, the standard approach includes the intraurethral administration of a local anesthetic or lubricant prior to the procedure to enhance patient comfort. While some patients tolerate the procedure well, others may exhibit heightened sensitivity and limited tolerance. Even in cases where the procedure is completed, the pain experienced and the resistance demonstrated by the patient may pose challenges for both the patient and the physician. Occasionally, a mismatch is observed between the patient's reported pain and the resistance displayed. The physician's perception of the patient's pain may also differ from the pain reported by the patient.

Previous studies have explored factors that can influence and reduce the perception of pain during cystoscopy performed under local anesthesia. However, data are lacking regarding the relationship between patients' pre-procedural anxiety and depression levels and the pain experienced during the procedure, as well as the physician's perception of that pain. The primary aim of the study is to compare the pain score reported by the patient with the pain level perceived by the physician. A secondary objective is to evaluate patients' pre-procedure anxiety and depression scores, along with their pain scores during the procedure, in the context of flexible cystoscopy performed under local anesthesia.

The study will include male patients aged 18 years and older who are undergoing cystoscopy due to urological complaints. Exclusion criteria include patients with known urethral strictures or those diagnosed with strictures during cystoscopy, individuals with allergies to the local anesthetic used, and patients with cardiopulmonary conditions that preclude the procedure.

Participants will be asked to complete the Hospital Anxiety and Depression Scale (HADS) for the assessment of general anxiety and depression, as well as the Visual Analog Scale (VAS) for pain and anxiety, at the time of admission. All patients will receive standard intraurethral local anesthesia 15 minutes prior to the procedure. Following cystoscopy, participants will complete the VAS for anxiety and pain again, 15 minutes after the procedure, to evaluate their intra-procedural experience. In addition, the physician performing the procedure will complete the VAS for anxiety and pain based on their perception of the patient's experience.

Patients will be randomized into four groups based on the experience level of the physician performing the procedure: a physician with more than five years of experience, a physician with less than five years of experience, a second-year resident under supervision, and a fourth-year resident. A total of 30 patients will be included in each group. The physician will remain blinded to the forms completed by the patient before and after the procedure and will independently assess the patient's condition.

ELIGIBILITY:
Minimum Age: 18 Years Maximum Age: Not Applicable Sex: Male Gender Based: Yes Male patients over 18 years of age who need cystoscopy due to urologic complaints will be included in the study.

Accepts Healthy Volunteers: No

Inclusion Criteria:

Male patients

Over 18 years of age

Patients for whom diagnostic cystoscopy is indicated for a urologic reason

Exclusion Criteria:

Female patients

Patients younger than 18 years of age

Patients with known urethral stricture

Patients with urethral stricture detected during cystoscopy

Patients who cannot tolerate flexible cystoscopy with local anesthesia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients over 18 years of age who need cystoscopy due to urologic complaints will be included in the study.
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Physicians' Perception about Patient Pain in Flexible Cystoscopy with Local Anesthesia | Immediately after the procedure, upon completion of the diagnostic flexible cystoscopy (15 minutes post-procedure).
  The study will examine the differences in the perception of pain scores in patients according to the years of experience of physicians.
  Scale Used: Visual Analog Scale (VAS) for Pain Minimum Value: 0 (No pain) Maximum Value: 10 (Worst possible pain) Interpretation: Higher scores indicate worse pain perception.

SECONDARY OUTCOMES:
Association between patients' pre-procedure HAD score and pain | Pre-procedure (baseline), immediately after the procedure (15 minutes post-procedure).
  Depression and anxiety levels in the pre-procedure HAD scores and VAS pain scores during the procedure will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Kamil Cam, Professor Doctor, Study Chair — Marmara University, School of Medicie, Department of Urology
Locations (1):
- Marmara University, School of Medicie, Department of Urology, Istanbul, Türkiye, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic data, Hospital Anxiety and Depression Scale (HADS) scores, and Visual Analog Scale (VAS) pain scores collected during the study will be shared with researchers upon request. The data will be anonymized to ensure participant privacy and confidentiality. The sharing will occur in compliance with ethical guidelines and institutional policies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available starting from the study completion date (September 15, 2025) and will be accessible for a period of 5 years.
Access Criteria: The IPD and supporting materials will be available to qualified researchers upon request. Researchers will have access to anonymized demographic data, Hospital Anxiety and Depression Scale (HADS) scores, Visual Analog Scale (VAS) pain scores, study protocol, statistical analysis plan, informed consent forms, and the final clinical study report. Access will be granted through a secure, password-protected data-sharing platform hosted by Marmara University, with adherence to ethical guidelines and confidentiality protocols. Requests can be made by contacting the study's central contact person, Dr. Gunal Ozgur (email: gunalozgur91@hotmail.com).
URL: https://www.marmarauroloji.com/

REFERENCES:
- [Background] Yeo JK, Cho DY, Oh MM, Park SS, Park MG. Listening to music during cystoscopy decreases anxiety, pain, and dissatisfaction in patients: a pilot randomized controlled trial. J Endourol. 2013 Apr;27(4):459-62. doi: 10.1089/end.2012.0222. Epub 2012 Dec 5. PMID 23009573
- [Background] Gezginci E, Bedir S, Ozcan C, Iyigun E. Does Watching a Relaxing Video During Cystoscopy Affect Pain and Anxiety Levels of Female Patients? A Randomized Controlled Trial. Pain Manag Nurs. 2021 Apr;22(2):214-219. doi: 10.1016/j.pmn.2020.08.005. Epub 2020 Sep 29. PMID 33008780
- [Background] Luczak M, Nowak L, Chorbinska J, Galik K, Kielb P, Laszkiewicz J, Tukiendorf A, Koscielska-Kasprzak K, Malkiewicz B, Zdrojowy R, Szydelko T, Krajewski W. Influence of Virtual Reality Devices on Pain and Anxiety in Patients Undergoing Cystoscopy Performed under Local Anaesthesia. J Pers Med. 2021 Nov 16;11(11):1214. doi: 10.3390/jpm11111214. PMID 34834565